CLINICAL TRIAL: NCT03857451
Title: Treatment of Gait Disorders in Children With Dravet Syndrome
Acronym: T-GaiD
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Ann Hallemans, Assistent Professor, Department of Rehabilitation Sciences and Physiotherapy, Faculty of Medicine and Health Science, Head of the Multidisciplinary Motor Center Antwerp, Universiteit Antwerpen
Other Study IDs: 34264; T003116N (Other Grant/Funding Number: Research Foundation - Flanders)
Record Dates: First submitted 2018-12-21; First posted 2019-02-28 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Dravet Syndrome; Severe Myoclonic Epilepsy of Infancy
Keywords: Dravet syndrome; severe myoclonic epilepsy of infancy; intellectual disabilities; movement disorders; gait; biomechanics
MeSH Terms: conditions — Epilepsies, Myoclonic; Intellectual Disability; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical gait analysis — Three dimensional gait analysis consisting of joint kinematics, kinetics and dynamic EMG data will be introduced into the diagnostic scheme

SUMMARY:
Dravet syndrome is a severe infantile onset epilepsy syndrome with a prevalence of 1/15.000 to 1/30.000. An infant with an apparently normal development presents around 6 months of age with a convulsive status epilepticus. Seizures can be triggered by fever, illness or vaccination. Because of its drug-resistance, in the past, most attention has been paid to seizure control. However, developmental and behavioural problems also become a serious concern during the second year of life. Outcome is poor, with intellectual disability and ongoing seizures. On the long term, the deterioration in gait is very characteristic. A crouch gait pattern develops that largely impacts the daily life functioning. Most children maintain the ability to walk around the house, but for longer distances they must rely on wheelchair use, which further negatively affects their mobility. Gait analysis, when combined with physical examination, provides quantitative information to guide treatment of gait disorders and assess its outcome. The goal of this project is the development of a clinical decision framework based upon 3D gait analysis to diagnose and treat mobility problems in children with Dravet syndrome. Two major university hospitals in Flanders (UZA and UZ Leuven) are partners in this project. The parent organisation "Stichting Dravetsyndroom Nederland/Vlaanderen" will also participate, as intermediate partner to facilitate contacts between all parties being patients and their caregivers, clinical gait labs and treating physicians.

DETAILED DESCRIPTION:
The problem under investigation is the reduced functional mobility of patients with Dravet syndrome resulting from a crouch gait pattern. The solution, proposed in this research project, is the development of a decision framework based upon clinical gait analysis to identify the main problems and subsequently use this knowledge to select the appropriate treatment for the observed gait disorder.

Dravet syndrome is a severe infantile onset epilepsy syndrome with a prevalence of 1/15.000 to 1/30.000. In 80% of the cases it is associated with mutations in the gene encoding the alpha-subunit of the sodium channel SCN1A that is expressed in the frontal lobe, basal ganglia and cerebellum. An infant with an apparently normal development presents around 6 months of age with a convulsive status epilepticus. Seizures can be triggered by fever, illness or vaccination. Because of its drug-resistance, in the past, most attention has been paid to seizure control. However, developmental and behavioural problems also become a serious concern during the second year of life. Outcome is poor, with intellectual disability and ongoing seizures. On the long term, the deterioration in gait is very characteristic. A crouch gait pattern develops that largely impacts the daily life functioning. Most children maintain the ability to walk around the house, but for longer distances they must rely on wheel-chair use, which further negatively affects their mobility. In general, Dravet syndrome is a very severe epileptic encephalopathy with a negative impact on the health and quality of life of both the patients and their caregivers.

Crouch gait refers to a sustained flexion of the hip, knee and ankle throughout the stance phase of gait. This is a very inefficient walking pattern with increased energy expenditure. Crouch gait is also observed in children with cerebral palsy (CP). In this population, ankle-foot orthoses (AFOs) show effective in resolving the underlying biomechanical deviations and improving functional mobility. Similar benefits can be expected in children with Dravet. However, before AFOs can be routinely applied in clinical practice, more research is necessary to identify the cause of crouch gait in patients with Dravet syndrome. The hypothesis was formulated that the crouch pattern in children with Dravet might develop as a consequence of lever arm dysfunctions in the lower limbs resulting from skeletal malalignment in combination with muscle weakness. The first objective in this study is to confirm this hypothesis. The second objective is to determine the effectiveness of AFOs in relieving the biomechanical problems, thereby reducing crouch gait and improving functional mobility. Pilot work in 10 children show primary problems situated around the ankle joint, providing proof of concept for the use of AFOs. In the first phase of the project, two research questions will be addressed.

1. Which biomechanical problems contribute to the crouch gait in children with Dravet syndrome?
2. Can AFO improve musculoskeletal alignment and reduce knee flexion in children with Dravet syndrome?

Gait analysis, when combined with physical examination, provides quantitative information to guide treatment of gait disorders and assess its outcome. At the University of Antwerp a state-of-the-art gait lab, the Multidisciplinary Motor Center Antwerp (M²OCEAN) was established in 2010 by means of a Hercules grant type 2 (AUHA/09/006). Since the Dravet consultation follows 80% of the children with Dravet syndrome in Flanders, the University of Antwerp is best placed to incorporate clinical gait analysis in the diagnostic scheme of these children. However, as a result of the mental retardation observed in these children, lengthy and time consuming protocols are a problem that can negatively affect the attainability of a good measurement. The mental retardation also becomes a problem when the children do not understand the instructions during physical examination. The challenge is to develop adequate protocols for both data collection and processing that specifically target the problems faced in this population. These protocols need to be feasible and understandable in children with low intelligence quotient. Information from the first phase of this project serves as input for this second phase that aims at answering the following questions:

1. Which protocols for clinical gait analysis are most suitable in children with Dravet syndrome?
2. What are the mobility benefits of applying the selected protocols for 3D gait analysis in clinical practice for children with Dravet syndrome? This project consists of 2 phases. The first phase (month 1 - 36) is directed at scientific research to validate the proof of concept for treatment of crouch gait in children with Dravet syndrome. The second phase (month 12 - 48) is dedicated to methodological developments that will enhance the routinely application of clinical gait analysis in the diagnostic scheme of children with Dravet syndrome and will provide proof that clinical gait analysis is a useful tool to identify main gait problems and set appropriate treatment goals in children with Dravet syndrome.

The overall design of choice for the first phase is a mixed longitudinal design. A cohort of children with Dravet syndrome will be subjected to follow-up for a period of 3 years annually receiving a physical examination and instrumented 3D clinical gait analyses (kinematics, kinetics, EMG). Two age-matched control groups will be retrospectively included. Control groups consist of a sample of age-matched typically developing children and a sample of age-matched children with cerebral palsy walking without and with AFO.

The work is organised into four work packages. The first work package (WP1) is dedicated to data collection and comprises the longitudinal follow up of the cohort of children with Dravet syndrome and the retrospective data collection in the control groups. Data will be collected throughout the first 3 years of the project. Case - control studies related to scientific goals 1 and 2 are organised in the second work package (WP2) whereby WP2.1 focusses on the identification of the biomechanical factors that contribute to the development of crouch gait and WP2.2 is directed at providing evidence that AFO can improve gait. The third work package (WP3) occurs synchronously in time and is related to the third research goal aiming at providing evidence for the benefit of including clinical gait analysis in the diagnostic scheme of children with Dravet syndrome. The last work package (WP4), the protocol selection and optimization, can start when the main biomechanical problems are identified in WP2.1.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Dravet syndrome according to the criteria of Ceulemans and Cras (2004)
* aged minimum 3 years and maximum 25 years at inclusion
* having minimum 1 year of walking experience

Exclusion Criteria:

* severe epileptic seizure (status epilepticus or tonic-clonic insult over 3 min) within the 24 hours before the assessment
* insufficient cooperation to perform 3D gait analysis
* comorbidities of other neurological and/or orthopedic disorders not linked to Dravet syndrome

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children and adolescents with Dravet syndrome living in Flanders and the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Lower limb kinematics during walking in degrees | baseline (at intake in year 1 of the study, T0)
  The gait pattern is assessed by instrumented 3D gait analysis using the standardized Vicon Clinical Gait Model. Joint rotation angles of the major joints of the lower limbs will be described during walking

SECONDARY OUTCOMES:
Lower limb kinematics during walking in degrees | after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  The gait pattern is assessed by instrumented 3D gait analysis using the standardized Vicon Clinical Gait Model. Joint rotation angles of the major joints of the lower limbs will be described during walking.
Lower limb kinetics during walking | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  The gait pattern is assessed by instrumented 3D gait analysis using the standardized Vicon Clinical Gait Model. Net forces acting around the major joints of the lower limbs will be calculated.
Muscle activation patterns during gait in microvolts | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Surface electromyography signals (microvolts) will be recorded during gait.
Functional strength on the Functional Strength Measurement. | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Functional muscle strength will be assessed during clinical examination using the Functional Strength Measurement (FSM). The FSM consists of eight items: overarm throwing (centimeters), chest pass (centimeters), standing long jump (centimeters), sit to stand (number of repetitions in 30 seconds), underarm throwing (centimeters), lifting a box (number of repetitions in 30 seconds), lateral step-up (numer of repetitions in 30 seconds) and stair climbing (number of steps in 30 seconds). Norm reference values are available.
Functional Mobility Scale | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Functional mobility will be assessed during parent interview using the Functional Mobility Scale (FMS). The FMS is a 6-point scale with maximum score of 6 being the most functional outcome (independent on all surfaces) and minimum score of 1 being the least functional outcome (uses wheelchair)
Mobility Questionnaire 28 | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Mobility limitations during daily activities inside and outside of the house will be assessed during parent interview using the validated Dutch translation of the Mobility Questionnaire 28 (MobQuest28), Dutch version: MobiliteitsVragenlijst 28 (MoVra28). The MobQuest28/MoVra28 consists of 28 items with a 5-point rating scale (0 = without any difficulties to 4 = impossible without help). A total score (0-100) indicates the mobility limitations.

OTHER OUTCOMES:
heigth in meters | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Total body height will be measured during clinical examination
body weigth in kilogram | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Body weight will be measured during clinical examination
passive joint range of motion in degrees | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Passive joint range of motion (°) will be measured during clinical examination using a goniometer
skeletal alignment in degrees | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Skeletal alignment will be measured during clinical examination using a goniometer
Muscle length in degrees | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  Hamstrings length (popliteal angle in degrees) and iliopsoas length (Thomas test in degrees) will be measured during clinical examination using a goniometer
Selective muscle strength on the Medical Research Council muscle scale | baseline (at intake in year 1 of the study, T0), after 12 months (T1), after 24 months (T2) and after 36 months (T3) from intake
  The Medical Research Council muscle scale is a 6-point scale with minimum score 0 = no muscle contraction and maximum score 5 = normal muscle power.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Hallemans, PhD, Principal Investigator — Rehabilitation Sciences and Physiotherapy, University of Antwerp
Locations (3):
- Belgium (3):
  - University Hospital Antwerp, Antwerp
  - University of Antwerp, Antwerp
  - KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Figueiredo EM, Ferreira GB, Maia Moreira RC, Kirkwood RN, Fetters L. Efficacy of ankle-foot orthoses on gait of children with cerebral palsy: systematic review of literature. Pediatr Phys Ther. 2008 Fall;20(3):207-23. doi: 10.1097/PEP.0b013e318181fb34. PMID 18703958
- [Background] Rodda JM, Scheffer IE, McMahon JM, Berkovic SF, Graham HK. Progressive gait deterioration in adolescents with Dravet syndrome. Arch Neurol. 2012 Jul;69(7):873-8. doi: 10.1001/archneurol.2011.3275. PMID 22409937
- [Background] Scheffer IE. Diagnosis and long-term course of Dravet syndrome. Eur J Paediatr Neurol. 2012 Sep;16 Suppl 1:S5-8. doi: 10.1016/j.ejpn.2012.04.007. Epub 2012 Jun 16. PMID 22704920
- [Result] Wyers L, Di Marco R, Zambelli S, Masiero S, Hallemans A, Van de Walle P, Desloovere K, Del Felice A. Foot-floor contact pattern in children and adults with Dravet Syndrome. Gait Posture. 2021 Feb;84:315-320. doi: 10.1016/j.gaitpost.2020.12.030. Epub 2021 Jan 6. PMID 33445140
- [Result] Verheyen K, Wyers L, Del Felice A, Schoonjans AS, Ceulemans B, Van de Walle P, Hallemans A. Independent walking and cognitive development in preschool children with Dravet syndrome. Dev Med Child Neurol. 2021 Apr;63(4):472-479. doi: 10.1111/dmcn.14738. Epub 2020 Nov 23. PMID 33230827
- [Result] Wyers L, Verheyen K, Ceulemans B, Schoonjans AS, Desloovere K, Van de Walle P, Hallemans A. Strength measurements in patients with Dravet Syndrome. Eur J Paediatr Neurol. 2021 Nov;35:100-110. doi: 10.1016/j.ejpn.2021.10.006. Epub 2021 Oct 15. PMID 34666230
- [Result] Wyers L, Verheyen K, Ceulemans B, Schoonjans AS, Desloovere K, Van de Walle P, Hallemans A. The mechanics behind gait problems in patients with Dravet Syndrome. Gait Posture. 2021 Feb;84:321-328. doi: 10.1016/j.gaitpost.2020.12.029. Epub 2020 Dec 31. PMID 33445141
- [Result] Wyers L, Van de Walle P, Hoornweg A, Tepes Bobescu I, Verheyen K, Ceulemans B, Schoonjans AS, Desloovere K, Hallemans A. Gait deviations in patients with dravet syndrome: A systematic review. Eur J Paediatr Neurol. 2019 May;23(3):357-367. doi: 10.1016/j.ejpn.2019.03.003. Epub 2019 Mar 22. PMID 30940509
- [Result] Di Marco R, Hallemans A, Bellon G, Ragona F, Piazza E, Granata T, Ceulemans B, Schoonjans AS, Van de Walle P, Darra F, Dalla Bernardina B, Vecchi M, Sawacha Z, Scarpa B, Masiero S, Benedetti MG, Del Felice A. Gait abnormalities in people with Dravet syndrome: A cross-sectional multi-center study. Eur J Paediatr Neurol. 2019 Nov;23(6):808-818. doi: 10.1016/j.ejpn.2019.09.010. Epub 2019 Sep 21. PMID 31582194
- [Result] Verheyen K, Verbecque E, Ceulemans B, Schoonjans AS, Van De Walle P, Hallemans A. Motor development in children with Dravet syndrome. Dev Med Child Neurol. 2019 Aug;61(8):950-956. doi: 10.1111/dmcn.14147. Epub 2019 Jan 15. PMID 30644536

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT03857451/Prot_001.pdf
  • Informed Consent Form (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03857451/ICF_000.pdf